CLINICAL TRIAL: NCT03844074
Title: A Clinical Effectiveness, Multicenter, Randomized, Double-masked, Controlled Study of the Efficacy and Safety of ONS-5010 in Subjects With Subfoveal Choroidal Neovascularization (CNV) Secondary to Age-related Macular Degeneration
Brief Title: A Clinical Effectiveness Study Examining the Efficacy and Safety of ONS-5010 in Subjects With Neovascular Age-related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Outlook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONS-5010-001
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Age-related Macular Degeneration; Neovascular Age-related Macular Degeneration; Wet Macular Degeneration
Keywords: Subfoveal Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bevacizumab (Experimental): ONS-5010
  Interventions: Biological: bevacizumab
- ranibizumab (Active Comparator)
  Interventions: Biological: ranibizumab

INTERVENTIONS:
Biological: bevacizumab — 1.25 mg, intravitreal injection
  Other Names: ONS-5010
  Arms: bevacizumab
Biological: ranibizumab — 0.5mg, intravitreal injection
  Arms: ranibizumab

SUMMARY:
This research study will examine the safety and effectiveness of ONS-5010 in participants with AMD. The goal is to prevent vision loss by evaluating the effectiveness of ONS-5010 as compared with ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* Active primary or recurrent Subfoveal Choroidal Neovascularization lesions secondary to Age-related macular degeneration (AMD) in the study eye
* Best corrected visual acuity of 20/40 to 20/320
* Study eye must:

  * Have active leakage on Fluorescein Angiogram involving the fovea
  * Have edema involving the fovea
  * Be free of foveal scarring
  * Be free of foveal atrophy

Exclusion Criteria:

* Previous use of anti-VEGF or bevacizumab within 6 weeks
* Previous subfoveal focal laser photocoagulation in the study eye
* Laser photocoagulation (juxtafoveal or extrafoveal) in the study eye within 1-month preceding randomization
* Any concurrent intraocular condition in the study eye that may require medical or surgical intervention or contribute to vision loss within 1 year
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous haemorrhage in the study eye
* Polypoidal choroidal vasculopathy (PCV) confirmed by indocyanine green angiography (ICGA)
* History of idiopathic or autoimmune-associated uveitis in either eye
* Infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥30 mmHg despite treatment with anti-glaucoma medication)
* Premenopausal women not using adequate contraception
* Current treatment for active systemic infection
* Known allergy to any component of the study drug or history of allergy to fluorescein or indocyanine green, not amenable to treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who gain 15 or more letters in the best corrected visual acuity (BCVA) score | Baseline, 11 months
  BCVA to be assessed as letters read using the Early Treatment Diabetic Retinopathy Study (ETDRS) charts. A positive change represents an improvement in visual acuity.

SECONDARY OUTCOMES:
Mean change in the best corrected visual acuity over time | Baseline, monthly to 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A positive change represents an improvement in visual acuity.
Proportion of participants who gain at least 10 letters in the best corrected visual acuity score | Baseline, 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A positive change represents an improvement in visual acuity.
Proportion of participants who gain at least 5 letters in the best corrected visual acuity score | Baseline, 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A positive change represents an improvement in visual acuity.
Proportion of participants who lose fewer than 15 letters in the best corrected visual acuity score | Baseline, 11 months
  BCVA to be assessed as letters read using the ETDRS charts. A negative change represents a decrease in visual acuity.
Proportion of participants with visual-acuity Snellen equivalent of 20/200 or worse | Baseline, 11 months
Percentage of participants with ocular adverse events, non-ocular adverse events, grade 3 and above laboratory abnormalities, and vital sign abnormalities | 11 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Kissner, PhD, Study Director — Outlook Therapeutics, Inc.
Locations (9):
- Australia (9):
  - Clinical Site, Hurstville, New South Wales
  - Clinical Site, Liverpool, New South Wales
  - Clinical Site, Sydney, New South Wales
  - Clinical Site, Westmead, New South Wales
  - Clinical Site, Brisbane, Queensland
  - Clinical Site, Adelaide, South Australia
  - Clinical Site, Hobart, Tasmania
  - Clinical Site, Essendon, Victoria
  - Clinical Site, Glen Waverley, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
Data will not be shared until all global regulatory filings are complete.